CLINICAL TRIAL: NCT00324558
Title: Multicenter, Randomized, Open and Sequential Study to Evaluate the Efficacy and Safety of Bemiparin Administration on the Response to Treatment in Patients Diagnosed With Limited Small Cell Lung Cancer
Brief Title: Adjuvant BEmiparin in Small Cell Lung Carcinoma (ABEL STUDY)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor stopped due to difficulties to recruit 130 patients required by protocol
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICT-BEM-2004-01; 2004-004722-27 (Nº EudraCT)
Record Dates: First submitted 2006-05-09; First posted 2006-05-11 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Carcinoma, Small Cell
Keywords: Bemiparin; small cell lung carcinoma
MeSH Terms: conditions — Carcinoma, Small Cell; Small Cell Lung Carcinoma | interventions — bemiparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Bemiparin 3,500 IU
  Interventions: Drug: Bemiparin
- Control (No Intervention)

INTERVENTIONS:
Drug: Bemiparin — subcutaneous administration (sc) of Bemiparin (3,500 UI/day) for 26 weeks, starting on the first day of chemotherapy (CT)
  Arms: 1

SUMMARY:
Main objective:

To evaluate whether the subcutaneous administration (sc) of Bemiparin (3,500 UI/day) for 26 weeks, starting on the first day of chemotherapy (CT), delays tumoral spread and increases progression-free survival.

Secondary objectives:

To evaluate whether the subcutaneous administration (sc) of Bemiparin (3,500 UI/day) for 26 weeks, starting with the onset of chemotherapy, increases global survival, improving the response rates to treatment with CT + RT (radiotherapy) and reduces the incidence of venous thromboembolism (VTE).

DETAILED DESCRIPTION:
There is clinical evidence indicative of the beneficial effects of heparin in the evolution of patients with cancer. Apart from the studies that in an indirect way demonstrated an increase in the survival of oncological patients who, because of presenting a venous thromboembolism episode, were treated with low molecular weight heparin (LMWH) in comparison with those treated with non-fractionated heparin; direct actions were also demonstrated from the use of heparin in the survival and tumour progression. The administration of LMWH together with Chemotherapy has been proved to increase the survival of patients diagnosed of cancer of the pancreas in relation to those only treated with chemotherapy. An increase in the global survival of advanced solid tumours, with no thromboembolic disease,has also been showed.

All this suggests that an improvement in the survival of patients is observed when heparin is added to the usual anti-tumour treatment, especially to those without spread disease, and this effect seems to be independent of the protection against the thromboembolic complications.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years old or older, of either sex, with a diagnosis of limited small cell lung cancer.
2. Patients with an ECOG functional state less than or equal to 2.
3. Informed consent to participate in the study.
4. Patients with a platelet count above 100,000/microlitre with no hemorrhagic symptomatology.

Exclusion Criteria:

1. Curative or palliative surgery as the initial treatment of their neoplastic condition.
2. Patients with an active hemorrhage in the past two months, organic lesions susceptible to bleeding (e.g. active peptic ulcer, hemorrhagic cerebrovascular accident, aneurysms), history of clinically evident hemorrhagic episodes, major surgery in the past month, outstanding clinically hemoptysis or an increased risk of bleeding due to any homeostatic alteration that contraindicates anticoagulant therapy.
3. Known hypersensitivity to LMWH, heparin or substances of porcine origin.
4. Patients with hypersensitivity to the chemotherapeutic agents used in this protocol that makes it impossible to use the antitumoral regime indicated in this protocol (cisplatin or carboplatin and etoposide), i.e. hypersensitivity to cisplatin and carboplatin or hypersensitivity to etoposide.
5. Patients with congenital or acquired bleeding diathesis.
6. Damage to/ or surgical interventions of the central nervous system, eyes and ears within the past 6 months.
7. Acute bacterial endocarditis or slow endocarditis.
8. Patients with a history of heparin-associated thrombocytopenia or with a current platelet count < 100,000/mm3
9. Patients with severe renal failure (serum creatinine over 2 mg/dl) or hepatic insufficiency (with values of AST and/or ALT > 5 times the normal value established in the reference range of the local hospital laboratory).
10. Severe arterial hypertension (systolic blood pressure over 200 mmHg and/or diastolic blood pressure above 120 mmHg).
11. Women who are pregnant or breast-feeding, or with the possibility of becoming pregnant during the study.
12. Patients with suspected inability/or inability to comply with treatment and/or complete the study.
13. Patients who are participating in another clinical trial or have done so in the past 30 days.
14. Patients with a life expectancy less than 3 months.
15. Patients on treatment with anticoagulants or who have been on treatment during three months before the diagnosis of the tumor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-06; Primary Completion 2010-02 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
efficacy: progression-free survival in months (measurements of the size of the effect will be done using the Kaplan Meier method and the difference between the means of this time) | efficacy
safety: will be the incidence, during randomized treatment period (from day 1 to the last day of treatment + 7 days), of major bleedings. | safety

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Gúrpide, MD, Principal Investigator — Clínica Universitaria de Navarra; Enrique Gonzalez, MD, Principal Investigator — Hospital General Universitario Morales Meseguer; Guillermo López, MD, Principal Investigator — Hopspital de Cruces, Baracaldo (Vizcaya); César Rodríguez, MD, Principal Investigator — Hospital Clínico de Salamanca; Juan C. Torrego, MD, Principal Investigator — Hospital del Rio Hortega; José Gómez, MD, Principal Investigator — Hospital La Fe de Valencia; Albert Font, MD, Principal Investigator — Germans Trias i Pujol Hospital; Isidoro C. Barneto, MD, Principal Investigator — Hospital Reina Sofia (Córdoba); Antonio Lorenzo, MD, Principal Investigator — Hospital de Puerto Real (Cádiz); Dolores Isla, MD, Principal Investigator — Hospital Clínico Lozano Blesa (Zaragoza); Eduardo Rocha, MD, Study Director — Clínica Universitaria de Navarra; Bartolomeu Massuti, MD, Principal Investigator — Hospital General Universitario de Alicante; Antonio Galán Brotons, MD, Principal Investigator — Hospital de Sagunto; Ana Blasco Cordellat, MD, Principal Investigator — Hospital General Universitario de Valencia; Juan J. Bretón, MD, Principal Investigator — Hospital Universitario Carlos Haya; Isabel Bover Barceló, MD, Principal Investigator — Hospital Son Llàtzer; Nuria Viñolas, MD, Principal Investigator — Hospital Clinic i provincial de Barcelona
Locations (15):
- Spain (15):
  - Hospital General de Alicante, Alicante, Alicante
  - Hospital Son Llàtzer, Son Ferriol, Balearic Islands
  - Hospital Clinic i Provicial de Barcelona, Barcelona, Barcelona
  - Hospital Clínico Universitario de Puerto Real, Puerto Real, Cádiz
  - Hospital Universitario Reina Sofía, Córdoba, Córdoba
  - Hospital Morales Meseguer, Murcia, Murcia
  - Hospital Universitario Carlos Haya, Málaga, Málaga
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - Hospital Clínico de Salamanca, Salamanca, Salamanca
  - Hospital de Sagunto, Port de Sagunt, Valencia
  - Hospital La Fe, Valencia, Valencia
  - Hospital General Universitario de Valencia, Valencia, Valencia
  - Hospital Río Hortega, Valladolid, Valladolid
  - Hospital de Cruces, Barakaldo, Vizcaya
  - Hospital Clínico Lozano Blesa, Zaragoza, Zaragoza

REFERENCES:
- [Derived] Rutjes AW, Porreca E, Candeloro M, Valeriani E, Di Nisio M. Primary prophylaxis for venous thromboembolism in ambulatory cancer patients receiving chemotherapy. Cochrane Database Syst Rev. 2020 Dec 18;12(12):CD008500. doi: 10.1002/14651858.CD008500.pub5. PMID 33337539
- [Derived] Lecumberri R, Lopez Vivanco G, Font A, Gonzalez Billalabeitia E, Gurpide A, Gomez Codina J, Isla D, Galan A, Bover I, Domine M, Vicente V, Rosell R, Rocha E. Adjuvant therapy with bemiparin in patients with limited-stage small cell lung cancer: results from the ABEL study. Thromb Res. 2013;132(6):666-70. doi: 10.1016/j.thromres.2013.09.026. Epub 2013 Sep 27. PMID 24491267